CLINICAL TRIAL: NCT00438568
Title: Therapeutic Effects of Intranasal Insulin Administration in AD
Brief Title: SNIFF 120: Study of Nasal Insulin to Fight Forgetfulness (120 Days)
Acronym: SNIFF 120
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30579-B; 5R01AG027415 (NIH); 1R01AG027415-01 (NIH)
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
Keywords: amyloid protein; brain metabolism; glucose metabolism; insulin sensitivity /resistance; cognition disorders
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Amyloidosis; Cognition Disorders | interventions — Insulin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): saline
  Interventions: Drug: Placebo
- 2 (Experimental): 10 Units
  Interventions: Drug: Regular Insulin
- 3 (Experimental): 20 Units
  Interventions: Drug: Regular Insulin

INTERVENTIONS:
Drug: Regular Insulin — administered intra-nasally twice a day for 16 weeks
  Other Names: Novolin U-100
  Arms: 2; 3
Drug: Placebo — administered intra-nasally twice a day for 16 weeks
  Other Names: saline
  Arms: 1

SUMMARY:
The purpose of this study is to find out if insulin, when administered as a "nasal spray" into the nasal passages, improves memory in adults with mild cognitive impairment (MCI) or Alzheimer's disease.

DETAILED DESCRIPTION:
A growing body of evidence suggests that insulin plays a role in normal memory processes and that insulin abnormalities may contribute to cognitive and brain changes associated with Alzheimer's disease (AD). Interestingly, insulin administered to the nasal cavity is transported within a few minutes into the brain, but does not affect blood sugar or insulin levels.

This study will consist of a randomized double-blind, placebo-controlled parallel group trial in which 90 participants with AD or MCI receive daily intranasal administrations of either insulin (10 or 20 IU twice a day for a total dose of 20 or 40 IU per day) or placebo (saline twice a day) for 4 months. The study will examine the effects of intranasal insulin administration on cognition, cerebral glucose metabolism, and β-amyloid (Aβ) in cerebrospinal fluid (CSF) and plasma, testing the hypothesis that daily intranasal insulin administration for 4 months will facilitate memory for adults with AD, and adults with mild cognitive impairment (MCI). A subset of participants will have the option to participate in 2 sub-studies: PET scans (prior to and at the end of treatment) to determine whether intranasal insulin increases cerebral glucose metabolism; lumbar punctures (LPs) before and at the end of treatment to determine effects of intranasal insulin administration on CSF Aβ levels.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 or greater
* Good physical health
* Memory impairment with a diagnosis of mild cognitive impairment (MCI) or Alzheimer's disease (AD)
* Participants on stable doses of Memantine (Namenda) or cholinesterase inhibitors will be eligible

Exclusion Criteria:

* Chronic sinus problems/allergies with chronic use of nasal decongestants or antihistamines
* Significant neurologic disease that might affect cognition (other than AD), such as stroke, Parkinson's disease, multiple sclerosis, severe head injury with loss of consciousness for more than 30 minutes or with permanent neurologic symptoms
* Significant medical illness or organ failure, such as uncontrolled hypertension or cardiovascular disease, chronic obstructive pulmonary disease, liver disease, or kidney disease
* Preexisting diabetes or current or previous use of hypoglycemic agents or insulin; participants will be excluded if they have a fasting blood sugar greater than 165 on baseline OGTT
* Clinically significant elevations in liver function tests, cholesterol, or triglycerides
* Major psychiatric disorders (e.g., untreated major depression and schizophrenia)
* Chronic use of the following types of medications: anti-psychotic, anxiolytic, and opiates

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2006-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Changes in cognition | every 8 weeks for 16 weeks, again at 8 weeks post-treatment (24 weeks)
glucose metabolism | every 8 weeks for 16 weeks, again at 8 weeks post-treatment (24 weeks)
plasma biological markers | every 8 weeks for 16 weeks, again at 8 weeks post-treatment (24 weeks)

SECONDARY OUTCOMES:
CSF biological markers | every 8 weeks for 16 weeks, again at 8 weeks post-treatment (24 weeks)
cerebral glucose metabolism | every 8 weeks for 16 weeks, again at 8 weeks post-treatment (24 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Principal Investigator — University of Washington
Locations (1):
- Veterans Administration Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Background] Reger MA, Watson GS, Frey WH 2nd, Baker LD, Cholerton B, Keeling ML, Belongia DA, Fishel MA, Plymate SR, Schellenberg GD, Cherrier MM, Craft S. Effects of intranasal insulin on cognition in memory-impaired older adults: modulation by APOE genotype. Neurobiol Aging. 2006 Mar;27(3):451-8. doi: 10.1016/j.neurobiolaging.2005.03.016. Epub 2005 Jun 16. PMID 15964100
- [Background] Reger MA, Craft S. Intranasal insulin administration: a method for dissociating central and peripheral effects of insulin. Drugs Today (Barc). 2006 Nov;42(11):729-39. doi: 10.1358/dot.2006.42.11.1007675. PMID 17171192
- [Background] Fishel MA, Watson GS, Montine TJ, Wang Q, Green PS, Kulstad JJ, Cook DG, Peskind ER, Baker LD, Goldgaber D, Nie W, Asthana S, Plymate SR, Schwartz MW, Craft S. Hyperinsulinemia provokes synchronous increases in central inflammation and beta-amyloid in normal adults. Arch Neurol. 2005 Oct;62(10):1539-44. doi: 10.1001/archneur.62.10.noc50112. PMID 16216936
- [Derived] Craft S, Baker LD, Montine TJ, Minoshima S, Watson GS, Claxton A, Arbuckle M, Callaghan M, Tsai E, Plymate SR, Green PS, Leverenz J, Cross D, Gerton B. Intranasal insulin therapy for Alzheimer disease and amnestic mild cognitive impairment: a pilot clinical trial. Arch Neurol. 2012 Jan;69(1):29-38. doi: 10.1001/archneurol.2011.233. Epub 2011 Sep 12. PMID 21911655